CLINICAL TRIAL: NCT00004441
Title: Study of Tauroursodeoxycholic Acid for Hepatobiliary Disease in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13439; CHMC-C-001439; CHMC-C-96-1-8; CHMC-C-FDR001439-01
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-07

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — ursodoxicoltaurine; Ursodeoxycholic Acid

INTERVENTIONS:
Drug: tauroursodeoxycholic acid
Drug: ursodiol

SUMMARY:
OBJECTIVES: I. Determine the optimum dose of tauroursodeoxycholic acid (TUDCA) required to achieve maximal bioavailability for patients with cystic fibrosis-associated liver disease.

II. Compare optimized doses of TUDCA with ursodiol (ursodeoxycholic acid; UDCA) for effects on biliary bile acid composition and metabolism, serum biochemistries, fat absorption, and fat-soluble vitamin status in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Objective I: This part of the study is a dose-response study to determine the optimal dose of tauroursodeoxycholic acid (TUDCA). Twenty-four patients are randomized to receive one of three different doses of TUDCA for 3 months.

Objective II: This part of the study is a double-blind crossover study to compare optimized doses of TUDCA with optimized doses of ursodiol in 15 patients stratified according to age (less than 10 vs 10-20 vs more than 20 years). Patients are randomized to receive either TUDCA or ursodiol orally for an initial 3 month period, followed by a 3 month washout period in which no drug is administered. Patients then receive the alternate drug for 3 months.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Cystic fibrosis-associated liver disease, defined by at least one of the following criteria: (1) Documented increase in serum concentrations of any of the liver enzymes (at least once in the preceding year) ALT at least twice normal AST at least 1.5 times normal Alkaline phosphatase at least 1.5 times normal GGT at least 1.5 times normal (2) Persistent hepatomegaly of more than 6 months duration defined by percussed liver span greater than 1 SEM for age (3) Splenomegaly, defined as a palpable spleen greater than 2.0 cm below the left costal margin (4) Abnormalities of ultrasound scan (increased size, dishomogeneous echogenicity, nodular liver, irregular margins, splenomegaly) within 6 months prior to study entry
* Patients enrolled in the first part of the study (objective I) are eligible to participate in the second part (objective II)

--Prior/Concurrent Therapy--

* At least 3 months since prior ursodiol
* At least 3 months since treatment with drug with choleretic properties or effects that influence bile acid metabolism

--Patient Characteristics--

* Hepatic: No decompensated cirrhosis No hepatic neoplasm or cholelithiasis
* Pulmonary: No significantly impaired pulmonary function with FEV1 less than 50%
* Other: At least 15 kg body weight No severely compromised clinical or nutritional state

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 1997-09; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Setchell, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (2):
  - Children's Hospital of Denver, Denver, Colorado
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
- University of Milan, Milan, Italy